CLINICAL TRIAL: NCT07330492
Title: Randomized Controlled Trial of a Nudge Intervention for Common Musculoskeletal Conditions
Brief Title: Testing a Brief Reassurance Message Before a Musculoskeletal Clinic Visit
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, David Ring, Associate Dean for Comprehensive Care; Professor and Associate Chair for Faculty Academic Affairs, Department of Surgery and Perioperative Care; Courtesy Professor of Psychiatry and Behavioral Sciences, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: STUDY00004831.3
Record Dates: First submitted 2025-12-15; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Any Non-traumatic Musculoskeletal Condition
Keywords: Musculoskeletal; Osteoarthritis; Nudge intervention; Behavioural intervention; Patient education; Healthcare utilization; Shared decision making; Reassurance
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Nudge / Reassurance Message) (Experimental): Participants randomized to the intervention group will read a brief, easy-to-understand message (generated by a Large Language Model) before their musculoskeletal clinic visit. The message explains that many musculoskeletal symptoms are common, often related to normal body changes, and can improve with simple self-care. It emphasizes that visits, tests, injections, and treatments are often optional, and patients can decide how much care they wish to pursue. After reading the message, participants will complete a short questionnaire rating their interest in follow-up visits, tests, injections, and surgery. Clinicians providing care will be blinded to participants' group assignment.
  Interventions: Behavioral: Nudge intervention
- Control arm (Usual Care) (No Intervention): Participants randomized to the control group will receive usual care prior to their musculoskeletal clinic visit, without any pre-visit reassurance message. They will complete the same questionnaire rating their interest in follow-up visits, tests, injections, and surgery. Clinicians providing care will be blinded to participants' group assignment.

INTERVENTIONS:
Behavioral: Nudge intervention — The intervention involves reading a brief, easy-to-understand message prior to a musculoskeletal clinic visit. The message explains that many musculoskeletal symptoms are common, often related to normal age-related changes, and can improve with simple self-care. It emphasizes that visits, tests, injections, and treatments are often optional, and patients can choose how much care to pursue.
  Other Names: Reassurance message
  Arms: Intervention Arm (Nudge / Reassurance Message)

SUMMARY:
The goal of this clinical trial is to learn if a brief, reassuring pre-visit message affects patients' expectations and planned follow-up care in adults with common musculoskeletal conditions. The main questions it aims to answer are:

* Does reading a brief reassurance message before a clinic visit change how interested patients are in additional care, such as follow-up visits, tests, injections, or surgery?
* Does the message affect whether patients actually schedule follow-up care after the visit?

Researchers will compare participants who receive the pre-visit reassurance message to those who receive usual care to see if the message changes patients' enthusiasm for care or their follow-up decisions.

Participants will:

1. Read a short, easy-to-understand message about musculoskeletal symptoms and options for care (for those in the intervention group)
2. Complete a brief questionnaire rating their interest in follow-up visits, tests, injections, or surgery
3. Have their scheduled follow-up care recorded after the clinic visit

ELIGIBILITY:
Inclusion Criteria:

* Adult (18+ years)
* English or Spanish language literacy
* Seeking musculoskeletal specialty care
* Diagnosed with any non-traumatic musculoskeletal condition
* New or return patient to clinic

Exclusion Criteria:

* Cognitive or other impairment precluding completion of a survey on a tablet
* Acute traumatic pathophysiology (fracture, dislocation, sprain/strain)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Pre-visit enthusiasm for additional care | Immediately after intervention
  The primary outcome is pre-visit enthusiasm for additional care, measured as participants' self-reported interest in pursuing a return visit, diagnostic tests, physical therapy, injections, or surgery. Participants rate each item on a 0-10 scale, where 0 indicates "not at all interested" and 10 indicates "definitely want it." This outcome is assessed immediately after the intervention (or usual care) and before the clinic visit.

SECONDARY OUTCOMES:
Actual scheduled follow-up care | Immediately following clinic visit
  The secondary outcomes are actual scheduled follow-up care after the musculoskeletal clinic visit, including return visits, diagnostic tests, physical therapy, injections, and surgery. These outcomes are recorded as yes/no for each type of care and are collected from the patient's medical record after the visit.

CONTACTS AND LOCATIONS:
Locations (1):
- Musculoskeletal Institute, UT Health Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-12-28): https://cdn.clinicaltrials.gov/large-docs/92/NCT07330492/Prot_SAP_000.pdf